CLINICAL TRIAL: NCT00040820
Title: A Treatment Access Program With Oxaliplatin for Previously Treated Colorectal Cancer Patients
Brief Title: Oxaliplatin in Treating Patients With Previously Treated Locally Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Miland Javle, MD, Roswell Park Cancer Institute
Purpose: Treatment
Other Study IDs: CDR0000069410; RPCI-DS-0130
Record Dates: First submitted 2002-07-08; First posted 2003-07-08 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Clinical trial to study the effectiveness of oxaliplatin in treating patients who have locally advanced or metastatic colorectal cancer that has been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide oxaliplatin for patients with previously treated locally advanced or metastatic colorectal cancer who have exhausted all approved therapies for colorectal cancer.

OUTLINE: This is a multicenter, Treatment Access Program study.

Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for at least 30 days.

PROJECTED ACCRUAL: Approximately one patient per site per month will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is not amenable to surgical resection or other potentially curative therapy

  * Locally advanced OR
  * Metastatic disease
* Patients who progressed on a non-oxaliplatin-containing (control) arm in Sanofi-Synthelabo second-line regulatory trials OR
* Patients who have exhausted all approved therapies for colorectal cancer (including fluorouracil and irinotecan) and have received at least 2 prior independent/different chemotherapy regimens
* Documented radiological disease progression after last anticancer treatment

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 75,000/mm3

Hepatic:

* SGOT or SGPT no greater than 6 times upper limit of normal (ULN)
* Bilirubin no greater than 2 mg/dL
* Alkaline phosphatase no greater than 5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* Adequate organ function and medically stable
* No known concurrent peripheral neuropathy
* Absence of deep tendon reflexes as the sole neurologic abnormality is allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 30 days since prior chemotherapy
* No prior oxaliplatin-based chemotherapy
* No other concurrent investigational chemotherapy agents

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 30 days since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 30 days since prior major surgical procedure or intervention

Other:

* At least 30 days since other prior anticancer therapy
* No other concurrent anticancer agents
* No concurrent participation in any other investigational studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2003-08 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States